CLINICAL TRIAL: NCT02487238
Title: A Single-Blind, Randomized, Placebo-Controlled Trial of Human Fecal Microbiota Transplantation for the Therapy of Pediatric Ulcerative Colitis and Inflammatory Bowel Disease Unclassified
Brief Title: Pediatric FEcal Microbiota Transplant for Ulcerative Colitis
Acronym: PediFETCh
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: McMaster Children's Hospital (Other)
Collaborators: London Health Sciences Centre (Other); St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Nikhil Pai, Assistant Professor, McMaster Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-364; NIF-15375 (Other Grant/Funding Number: Hamilton Health Sciences New Investigator Fund 2015); HAH-17-002 (Other Grant/Funding Number: AHSC AFP Innovation Fund 2016-2017)
Record Dates: First submitted 2015-06-25; First posted 2015-07-01 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Inflammatory Bowel Disease; Ulcerative Colitis
Keywords: Microbiome; Microbiota; Fecal Microbial Transplant; Fecal Microbiota Transplant; FMT; Gastroenterology; IBD; Inflammatory Bowel Disease; Ulcerative Colitis; UC; Inflammatory Bowel Disease Unclassified; IBD-U; Rebiotix; RBX2660; Pediatrics; McMaster Children's Hospital; Centre Hospitalier Universitaire Sainte-Justine; Children's Hospital at London Health Sciences Centre
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to receive either the fecal microbial enema containing healthy donor stool OR the normal saline enema placebo. Patients who receive the normal saline enema placebo may be eligible to still receive the fecal microbial enema when they finish the trial.
Who Masked: Participant
Masking Description: Patients will not be aware of which type of enema they have been randomized to receive (fecal microbial enema, or normal saline enema). Patients who were randomized to the normal saline enema will still be eligible to receive the fecal microbial enema when they finish the trial; these patients will know what they are receiving and no longer need masking.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fecal Microbiota Enema (Experimental): Live, healthy, human donor stool prepared as fecal enemas. Fecal enemas are prepared and collected by Rebiotix(®) (RBX2660), using extensively screened donor stool. Enemas will be administered on site at one of the participating trial sites by trained study investigators. Enemas are given: 2x per week for 6 weeks (total = 12 enemas over 6 weeks). Patients will be masked to enema contents.
  Interventions: Biological: Fecal Microbiota Enema
- Normal Saline Enema (Placebo Comparator): Normal saline enemas will be administered on site at one of the participating trial sites by trained study investigators. Enemas are given: 2x per week for 6 weeks (total = 12 enemas over 6 weeks). Patients will be masked to enema contents.
  Interventions: Biological: Normal Saline Enema

INTERVENTIONS:
Biological: Fecal Microbiota Enema — Active intervention.
  Other Names: FMT; RBX2660; Rebiotix; Fecal microbial enema
  Arms: Fecal Microbiota Enema
Biological: Normal Saline Enema — Placebo comparator.
  Arms: Normal Saline Enema

SUMMARY:
The PediFETCh study is a pilot trial designed to assess the feasibility of fecal microbiota transplants for the therapy of pediatric ulcerative colitis (UC) and pediatric inflammatory bowel disease-unclassified (IBD-U). Investigators will test the hypothesis that a protocol of twice-weekly retention enemas delivered over six weeks, using fecal transplant material from a healthy donor, will improve clinical and biological disease markers in patients with pediatric UC or IBD-U.

DETAILED DESCRIPTION:
BACKGROUND:

Approximately 104,000 Canadians are affected by ulcerative colitis (UC), an inflammatory bowel disease characterized by immune dysregulation. Ontario, Canada has some of the highest rates of childhood-onset UC in the world and this disease can be particularly debilitating in childhood. Effects on growth and development are profound in pediatric onset disease, and existing treatments, which include long-term immunosuppression, carry short and long-term risks of infection, malignancy, and toxicity.

The intestinal bacteria has a critical role in the regulation of the immune system. Fecal microbiota transplantation (FMT), the transfer of intestinal bacteria from a healthy donor to a recipient, has been shown to treat recurrent Clostridium difficile intestinal infections. The therapeutic potential of FMT for UC has been demonstrated in a recent adult UC trial at our institution (primary investigator: Dr. Paul Moayyedi; collaborator on the PediFETCh trial). Randomized, placebo-controlled trials of FMT in pediatric inflammatory bowel disease are nonexistent. FMT may present a valuable, safer therapeutic option for pediatric UC and a randomized-controlled trial is needed.

Four small case-series have demonstrated success of FMT for pediatric inflammatory bowel disease (IBD). Protocols and response rates varied across each study, but lower gastrointestinal tract administration yielded clinical response rates in 67-100% of patients. Two single--center pediatric case reports have been recently published showing marked clinical improvement in two patients with severe colitis. A 2015 case report described an 18 -month old female presenting with an early -onset colitis with UC- like presentation. She responded after 7 serial FMT infusions with donor stool from an age-matched niece and older brother. A 2016 case report described an 11 -year old female with steroid dependent UC who responded after serial FMT infusions every 2 to 4 weeks over a 10 month period. The patient remained in clinical remission at 40 weeks post final FMT, and showed complete endoscopic healing. A further 2016 case report described a 3-year old female with acute severe UC who was refractory to aminosalicylates and all immunosuppressive drugs. She received 6 successive FMT enemas and 4 FMT via nasoduodenal tube over 10 days. While this patient ultimately required colectomy, she did not show any significant long-term side effects as a result of the trial of FMT.

Strong evidence exists in adult studies to support the use of FMT in UC treatment. Four randomized-controlled trials (RCTs), considered one of the highest qualities of clinical trial evidence, have been published to date. Slight variations in protocol existed across all four studies, but taken together, the overall clinical and endoscopic remission rates in patients who received FMT were an impressive: 42.1% and 26.4%, respectively.

OBJECTIVES:

Our objective is to determine whether FMT can improve clinical, biological, and mucosal disease status in pediatric UC and IBD Unclassified (IBD-U). This pilot study will provide access to FMT treatment and demonstrate the feasibility of our study design in order to establish a framework for future studies for assessing the effectiveness of FMT intervention.

HYPOTHESES:

Based on previously published case series in pediatrics, single-patient case reports, and a recent randomized controlled trial in adults, we hypothesize that patients receiving fecal microbiota enemas containing healthy donor bacteria will experience clinical remission, improvement in inflammatory markers, and a longer duration of remission compared to patients receiving the placebo.

STUDY DESIGN:

The proposed study is a multicenter, randomized, controlled, single-blind trial. Pediatric patients with a diagnosis of UC, or IBD-U will be enrolled and randomized to receive 6 weeks of bi-weekly fecal microbiota enemas or normal saline enemas (placebo). Fecal enemas will contain healthy donor stool that has been extensively safety-screened and provided by Rebiotix® (RBX-2660).

Patients may continue taking their existing UC medical treatments (probiotics, 5-ASAs, immunomodulators, anti-TNF) while enrolled in the trial. However, no significant changes in dosing or the introduction of new therapies will be permitted over the study period. All fecal enemas will be delivered at the study site by investigators to ensure consistency in technique and viability of fecal transplant material. Patients will have clinical disease activity scores measured at each enema administration (6 weeks), and at weeks 18 and 30. Stool samples will be collected at time points throughout the trial for microbiome analyses and fecal calprotectin measurements, with support from the Farncombe Family Digestive Health Research Institute. Bloodwork will be collected throughout the trial to further measure change in biological disease activity.

Patients participating in the trial will be offered an opportunity to be re-enrolled in the fecal microbiota arm if they were initially randomized to the normal saline (placebo) arm of the study.

SAMPLE SIZE:

50 patients will be recruited for the trial across all participating study sites. Patients will be single-blinded, and randomized to placebo or treatment arms.

SAFETY MONITORING:

Study risks include complications of fecal microbiota transplants (infection, mild gastrointestinal symptoms, fever). Based on results of previous studies, and existing safety data of the fecal enema preparation (RBX2660) from previously conducted trials, the risks of infection, adverse gastrointestinal symptoms, or other adverse events are extremely low. The fecal enema preparation used in this trial (RBX2660) by Rebiotix(®) has received FDA IND and Health Canada approvals for clinical trials in recurrent C. difficile. Donors are initially prescreened, and donor blood and stool are extensively screened at additional time points prior to administration. We will be providing close follow-up of our patients throughout the trial and in followup.

OUTCOMES:

1. Primary outcomes for this pilot trial are measures of feasibility.
2. Secondary outcomes are measures of clinical response to fecal microbiota transplant treatments. These include: clinical response (based on Pediatric Ulcerative Colitis Activity Index [PUCAI] scores), biological response (serum bloodwork measures), mucosal healing (fecal calprotectin levels), and change in fecal microbiome (change in 16s rRNA, inferred metagenome, metabolome). Patients enrolled in the open-label portion of the trial will also have urine metabolomics measured. We will not be assessing other indices of mucosal healing, such as performing endoscopy or magnetic resonance enterography in this trial.

ELIGIBILITY:
Inclusion Criteria:

* 3yo to 17yo at start of trial
* Followed at a participating clinical trial site: a) McMaster Children's Hospital, b) Children's Hospital at London Health Sciences Centre, c) Centre Hospitalier Universitaire Sainte-Justine
* Ulcerative colitis (UC) or Inflammatory bowel disease unclassified (IBD-U)
* Evidence of active clinical, biological, or mucosal disease
* Ongoing treatment is acceptable provided the patient has had no significant changes to medications, or medication dose for at least 4 weeks prior to starting the trial

Exclusion Criteria:

* Active participation in another therapeutic trial
* Unable to give informed consent, or assent
* Active Clostridium difficile infection
* Significant change in medication type, or medication dose within the preceding 4 weeks prior to starting the trial
* Starting new treatments, or having a significant change in medication dosing during the trial
* Significant, consecutive rise in PUCAI score during the trial
* Hospitalization during trial

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2015-11; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Feasibility (Composite Measure) | 30 weeks
  Evaluation of: participant recruitment/retention/eligibility/acceptance/adverse events

SECONDARY OUTCOMES:
Microbiome Change (Composite Measure) | Weeks: 0/3/6/12/18/24/30
  Change in microbial community structure/inferred metagenomic/metabolome
Clinical Remission | Weeks: 0/1/2/3/4/5/6/12/18/24/30
  PUCAI score <10
Clinical Improvement | Weeks: 0/1/2/3/4/5/6/12/18/24/30
  Decrease in PUCAI score
Biological Improvement | Weeks: 0/3/6/18/30
  Decrease in ESR/C-reactive protein, Increase in hemoglobin/albumin
Mucosal Healing | Weeks: 0/3/6/12/18/24/30
  Decrease in fecal calprotectin
Urine Metabolomics Change | Weeks: 0/3/6/12/18/24/30
  Change in urine metabolomics profile (Open Label arm only)

CONTACTS AND LOCATIONS:
Overall Officials: Nikhil Pai, MD FRCPC, Principal Investigator — McMaster Children's Hospital; Jelena Popov, BSc, Study Director — McMaster Children's Hospital Division of Pediatric Gastroenterology & Nutrition; Tim Ramsay, PhD, Study Chair — The Ottawa Hospital Research Institute
Locations (3):
- Canada (3):
  - McMaster Children's Hospital, Hamilton, Ontario
  - Children's Hospital London Health Science Centre, London, Ontario
  - CHU Sainte-Justine, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Protocol has been published in BMJ Protocols 2017.
Supporting Information: Study Protocol, SAP
Time Frame: Open-access.
Access Criteria: Pai N, Popov J. Protocol for a randomised, placebo-controlled pilot study for assessing feasibility and efficacy of faecal microbiota transplantation in a paediatric ulcerative colitis population: PediFETCh trial. BMJ Open. 2017;7(8):e016698.
URL: http://bmjopen.bmj.com/content/7/8/e016698

REFERENCES:
- [Background] Rossen NG, Fuentes S, van der Spek MJ, Tijssen JG, Hartman JH, Duflou A, Lowenberg M, van den Brink GR, Mathus-Vliegen EM, de Vos WM, Zoetendal EG, D'Haens GR, Ponsioen CY. Findings From a Randomized Controlled Trial of Fecal Transplantation for Patients With Ulcerative Colitis. Gastroenterology. 2015 Jul;149(1):110-118.e4. doi: 10.1053/j.gastro.2015.03.045. Epub 2015 Mar 30. PMID 25836986
- [Background] Moayyedi P, Surette MG, Kim PT, Libertucci J, Wolfe M, Onischi C, Armstrong D, Marshall JK, Kassam Z, Reinisch W, Lee CH. Fecal Microbiota Transplantation Induces Remission in Patients With Active Ulcerative Colitis in a Randomized Controlled Trial. Gastroenterology. 2015 Jul;149(1):102-109.e6. doi: 10.1053/j.gastro.2015.04.001. Epub 2015 Apr 7. PMID 25857665
- [Background] Michail S, Durbin M, Turner D, Griffiths AM, Mack DR, Hyams J, Leleiko N, Kenche H, Stolfi A, Wine E. Alterations in the gut microbiome of children with severe ulcerative colitis. Inflamm Bowel Dis. 2012 Oct;18(10):1799-808. doi: 10.1002/ibd.22860. Epub 2011 Dec 14. PMID 22170749
- [Background] Kunde S, Pham A, Bonczyk S, Crumb T, Duba M, Conrad H Jr, Cloney D, Kugathasan S. Safety, tolerability, and clinical response after fecal transplantation in children and young adults with ulcerative colitis. J Pediatr Gastroenterol Nutr. 2013 Jun;56(6):597-601. doi: 10.1097/MPG.0b013e318292fa0d. PMID 23542823
- [Background] Kellermayer R, Nagy-Szakal D, Harris RA, Luna RA, Pitashny M, Schady D, Mir SA, Lopez ME, Gilger MA, Belmont J, Hollister EB, Versalovic J. Serial fecal microbiota transplantation alters mucosal gene expression in pediatric ulcerative colitis. Am J Gastroenterol. 2015 Apr;110(4):604-6. doi: 10.1038/ajg.2015.19. No abstract available. PMID 25853207
- [Background] Suskind DL, Brittnacher MJ, Wahbeh G, Shaffer ML, Hayden HS, Qin X, Singh N, Damman CJ, Hager KR, Nielson H, Miller SI. Fecal microbial transplant effect on clinical outcomes and fecal microbiome in active Crohn's disease. Inflamm Bowel Dis. 2015 Mar;21(3):556-63. doi: 10.1097/MIB.0000000000000307. PMID 25647155
- [Background] Vandenplas Y, Veereman G, van der Werff Ten Bosch J, Goossens A, Pierard D, Samsom JN, Escher JC. Fecal Microbial Transplantation in Early-Onset Colitis: Caution Advised. J Pediatr Gastroenterol Nutr. 2015 Sep;61(3):e12-4. doi: 10.1097/MPG.0000000000000281. No abstract available. PMID 24399213
- [Background] Shimizu H, Arai K, Abe J, Nakabayashi K, Yoshioka T, Hosoi K, Kuroda M. Repeated fecal microbiota transplantation in a child with ulcerative colitis. Pediatr Int. 2016 Aug;58(8):781-5. doi: 10.1111/ped.12967. Epub 2016 Jun 21. PMID 27324973
- [Background] Kumagai H, Yokoyama K, Imagawa T, Inoue S, Tulyeu J, Tanaka M, Yamagata T. Failure of Fecal Microbiota Transplantation in a Three-Year-Old Child with Severe Refractory Ulcerative Colitis. Pediatr Gastroenterol Hepatol Nutr. 2016 Sep;19(3):214-220. doi: 10.5223/pghn.2016.19.3.214. Epub 2016 Sep 29. PMID 27738605
- [Background] Narula N, Kassam Z, Yuan Y, Colombel JF, Ponsioen C, Reinisch W, Moayyedi P. Systematic Review and Meta-analysis: Fecal Microbiota Transplantation for Treatment of Active Ulcerative Colitis. Inflamm Bowel Dis. 2017 Oct;23(10):1702-1709. doi: 10.1097/MIB.0000000000001228. PMID 28906291
- [Background] Suskind DL, Singh N, Nielson H, Wahbeh G. Fecal microbial transplant via nasogastric tube for active pediatric ulcerative colitis. J Pediatr Gastroenterol Nutr. 2015 Jan;60(1):27-9. doi: 10.1097/MPG.0000000000000544. PMID 25162366
- [Background] Paramsothy S, Kamm MA, Kaakoush NO, Walsh AJ, van den Bogaerde J, Samuel D, Leong RWL, Connor S, Ng W, Paramsothy R, Xuan W, Lin E, Mitchell HM, Borody TJ. Multidonor intensive faecal microbiota transplantation for active ulcerative colitis: a randomised placebo-controlled trial. Lancet. 2017 Mar 25;389(10075):1218-1228. doi: 10.1016/S0140-6736(17)30182-4. Epub 2017 Feb 15. PMID 28214091
- [Background] Wang AY, Popov J, Pai N. Fecal microbial transplant for the treatment of pediatric inflammatory bowel disease. World J Gastroenterol. 2016 Dec 21;22(47):10304-10315. doi: 10.3748/wjg.v22.i47.10304. PMID 28058011
- [Background] Cammarota G, Ianiro G, Tilg H, Rajilic-Stojanovic M, Kump P, Satokari R, Sokol H, Arkkila P, Pintus C, Hart A, Segal J, Aloi M, Masucci L, Molinaro A, Scaldaferri F, Gasbarrini G, Lopez-Sanroman A, Link A, de Groot P, de Vos WM, Hogenauer C, Malfertheiner P, Mattila E, Milosavljevic T, Nieuwdorp M, Sanguinetti M, Simren M, Gasbarrini A; European FMT Working Group. European consensus conference on faecal microbiota transplantation in clinical practice. Gut. 2017 Apr;66(4):569-580. doi: 10.1136/gutjnl-2016-313017. Epub 2017 Jan 13. PMID 28087657
- [Background] Costello SP, Waters O, Bryant RV, et al. Short Duration, Low Intensity, Pooled Fecal Microbiota Transplantation Induces Remission in Patients with Mild-Moderately Active Ulcerative Colitis: A Randomised Controlled Trial. Gastroenterology 152(5): S198-S199, 2017.
- [Result] Pai N, Popov J. Protocol for a randomised, placebo-controlled pilot study for assessing feasibility and efficacy of faecal microbiota transplantation in a paediatric ulcerative colitis population: PediFETCh trial. BMJ Open. 2017 Aug 21;7(8):e016698. doi: 10.1136/bmjopen-2017-016698. PMID 28827258
- See also: Protocol for a randomised, placebo-controlled pilot study for assessing feasibility and efficacy of faecal microbiota transplantation in a paediatric ulcerative colitis population: PediFETCh trial — http://bmjopen.bmj.com/content/7/8/e016698